CLINICAL TRIAL: NCT02827929
Title: Efficacy of Education Programs in Patients With Chronic Airway Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Kwang-Ha Yoo, Professor, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ESR-14-10193
Record Dates: First submitted 2016-06-29; First posted 2016-07-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- educated group (Experimental): Subjects who is diagnosed as COPD or asthma by their physicians were recruited from 43 primary clinic and had been visiting each primary clinic over one year or more will be provided education of 3 times for one months about disease, inhaler use technics and action plans about exacerbation
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — 3 times systemic education program will be provided to patients were diagnosed as asthma or COPD by their physicians.

SUMMARY:
The objective of this study is to determine whether the systematic education on air way disease and inhalers in outpatient settings contributes to improve the quality of life.

Education has been known to be effective for management of chronic airway disease. However, the real benefits remain unclear. An organized education on the chronic airway disease is directed by primary care physicians, and the investigators evaluate the effectiveness of the education.

DETAILED DESCRIPTION:
The present study is a prospective and interventional study comparing the outcomes of education program for one month.

A one month education program is composed of three visits (every two weeks follow-up ) during which subjects were taught about their diseases, action plans in acute exacerbation, and inhaler technique.

To evaluate the effectiveness of systematic education, questionnaires evaluating quality of life and satisfaction of education will be examined after each visit.

Asthma control test (ACT) in asthma, chronic obstructive pulmonary disease (COPD) assessment test (CAT) in COPD subjects were compared before and after education as an index of quality of life.

Educational effects were also measured, associated with improvement of their knowledge for chronic airway disease itself, proper use of inhaler technique, and satisfaction of subjects after education.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as asthma or COPD
2. Patients of over 20 years old
3. Patients who agree with voluntary informed consent
4. Patients who were prescribed inhaler medication as treatment option

Exclusion Criteria:

1. Patients who have comorbid disorders which can influence on the study result (e.g. severe cardiac or kidney disease, cancer, transplantation, bronchiectasis, tuberculous destroyed lung)
2. Pregnant women
3. Patients who refused to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2014-06; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in CAT score | one month
  The investigators examined change of quality of life through CAT in patient with COPD.

SECONDARY OUTCOMES:
Change in ACT score | one month
  The investigators examined change of quality of life through Asthma control test in patient with asthma.
Medical cost | one month
  The investigators will compare the total medical cost related COPD or asthma before education with that after education. (unit: Korean won, KRW)
Compliance to Medication | one month
  Compliance is calculated as the ratio between the number of actual doses and the number of doses that should have been taken during the total treatment period. The investigators will compare the ratio before and after education about air way disease
patients satisfaction score with the education program | one month
physicians satisfaction score with the education program | one month
the time of acute exacerbation | one month

CONTACTS AND LOCATIONS:
Overall Officials: Kwang-Ha NA Yoo, M.D, Principal Investigator — Konkuk University Hospial
Locations (1):
- Konkuk University Hospital, Gwangjin-gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valero C, Monteagudo M, Llagostera M, Bayona X, Granollers S, Acedo M, Ferro JJ, Rodriguez-Latre L, Almeda J, Munoz L; COPD Group of SAP Baix LLobregat Centre. Evaluation of a combined strategy directed towards health-care professionals and patients with chronic obstructive pulmonary disease (COPD): information and health education feedback for improving clinical monitoring and quality-of-life. BMC Public Health. 2009 Dec 1;9:442. doi: 10.1186/1471-2458-9-442. PMID 20128887
- [Background] Wacker ME, Jorres RA, Karch A, Wilke S, Heinrich J, Karrasch S, Koch A, Schulz H, Watz H, Leidl R, Vogelmeier C, Holle R; COSYCONET-Consortium. Assessing health-related quality of life in COPD: comparing generic and disease-specific instruments with focus on comorbidities. BMC Pulm Med. 2016 May 10;16(1):70. doi: 10.1186/s12890-016-0238-9. PMID 27160582
- [Background] Koblizek V, Novotna B, Zbozinkova Z, Hejduk K. Diagnosing COPD: advances in training and practice - a systematic review. Adv Med Educ Pract. 2016 Apr 4;7:219-31. doi: 10.2147/AMEP.S76976. eCollection 2016. PMID 27099544
- [Background] Leiva-Fernandez J, Vazquez-Alarcon RL, Aguiar-Leiva V, Lobnig-Becerra M, Leiva-Fernandez F, Barnestein-Fonseca P. Efficacy of an educational intervention in primary health care in inhalation techniques: study protocol for a pragmatic cluster randomised controlled trial. Trials. 2016 Mar 17;17(1):144. doi: 10.1186/s13063-016-1269-5. PMID 26988095